CLINICAL TRIAL: NCT05052229
Title: Pulmonary Gas Exchange and Neuro-sensory Abnormalities in Patients With Idiopathic Pulmonary Fibrosis and Mild Mechanical Restriction. Implications for Dyspnea and Exercise Intolerance
Brief Title: Inhaled Nitric Oxide (iNO) in Idiopathic Pulmonary Fibrosis (IPF).
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Dr. Denis O'Donnell (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor-Investigator, Dr. Denis O'Donnell, Principal Investigator, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: DMED 2495-21; BI 1199.0477 (Other Grant/Funding Number: Boehringer Ingelheim Canada)
Record Dates: First submitted 2021-09-02; First posted 2021-09-22 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Exertional Dyspnea; Exercise; Nitric Oxide; Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Motor Activity | interventions — Nitric Oxide; Air

STUDY DESIGN:
Intervention Model Description: Single center, randomized, double-blind, cross-over design
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Inhaled medical grade normoxic gas (FiO2 = 0.21; DIN 02238755 Air Liquide Healthcare, Montreal, Quebec, Canada).
  Interventions: Drug: Medical air
- Nitric Oxide (Active Comparator): Inhaled 40 ppm nitric oxide from a KINOX gas cylinder system (Air Liquid Healthcare, Montreal, Quebec, Canada; DIN 02451328).
  Interventions: Drug: Nitric Oxide

INTERVENTIONS:
Drug: Nitric Oxide — Nitric oxide gas for inhalation
  Other Names: KINOX
  Arms: Nitric Oxide
Drug: Medical air — Medical grade air for inhalation (placebo)
  Other Names: Medical grade air
  Arms: Placebo

SUMMARY:
Idiopathic Pulmonary Fibrosis (IPF) is a progressive lung disease marked by reduced exercise capacity and activity-related breathlessness (commonly termed dyspnea). Our previous work has shown that dyspnea during exercise is associated with an increased drive to breathe (inspiratory neural drive; IND). However, little work has been done to understand the mechanisms of exertional dyspnea in patients with mild IPF. The objectives of this study are to compare the acute effects of inhaled nitric oxide to placebo on ventilatory efficiency (VE/VCO2), and IND at rest and during a standard cardiopulmonary exercise test (CPET). Twenty patients with diagnosed IPF with mild (or absent) mechanical restriction and 20 healthy age- and sex-matched controls will be recruited from a database of volunteers and from the Interstitial Lung Disease and Respirology clinics at Hotel Dieu Hospital. Participants with cardiovascular, or any other condition that contributes to dyspnea or abnormal cardiopulmonary responses to exercise will be excluded. After giving written informed consent, all participants will complete 7 visits, conducted 2 to 7 days apart. Visit 1 (screening): medical history, pulmonary function testing and a symptom limited incremental CPET. Visit 2: Standard CT examination conducted at KGH Imaging. Visit 3: assessment of resting chemoreceptor sensitivity, followed by a symptom limited incremental CPET to determine peak work rate (Wmax). Visits 4 & 5 (run-in): familiarization to standardized constant work rate (CWR) CPET to symptom limitation at 75% Wmax. Visits 6 & 7 (Randomized & Blinded): CWR CPET to symptom limitation while breathing a gas mixture with either 1) 40 ppm iNO or 2) placebo [medical grade normoxic gas, 21% oxygen]. The proposed work has the potential to provide important physiological insights into the underlying mechanisms of heightened dyspnea, as well as examine therapeutic avenues to improve quality of life in patients with IPF.

DETAILED DESCRIPTION:
Idiopathic pulmonary fibrosis (IPF) is a progressive fibrotic interstitial lung disease characterized by bi-basilar sub-pleural honeycombing, septal thickening, and traction bronchiectasis. Patients with IPF, even in mild cases, have a reduced exercise capacity which is strongly associated with exertional breathlessness (dyspnea). Our previous work in IPF has shown that dyspnea during exercise is associated with increased inspiratory neural drive (IND) compared with healthy controls. High IND, in turn, is related to a combination of 1) reduced ventilatory efficiency (i.e. increased ventilation relative to carbon dioxide production (V̇E/V̇CO2)); 2) abnormal dynamic breathing mechanics (blunted tidal volume (VT) and critically low inspiratory reserve volume (IRV)), especially in more advanced disease, and; 3) impaired pulmonary gas-exchange (i.e. diffusion limitation and arterial hypoxemia).

Preliminary work from our laboratory in patients with IPF but only mild restriction (total lung capacity (TLC) >70% predicted) demonstrated elevated IND and dyspnea during exercise, when compared to healthy age- and sex-matched controls. The increased IND appeared to be largely the result of the excess ventilation (high V̇E/V̇CO2), as dynamic respiratory mechanics (VT and operating lung volumes) during exercise were similar to healthy controls, when accounting for ventilation. Importantly, these patients showed only minor decreases in arterial O2 saturation. These data suggest that patients with mild forms of IPF have significant exertional dyspnea, secondary to reduced ventilatory efficiency (high V̇E/V̇CO2), although the exact mechanisms of elevated V̇E/V̇CO2 in mild IPF remains unclear.

Increased chemosensitivity has been linked to elevated V̇E/V̇CO2 in cardiopulmonary diseases. It is reasonable to postulate that persistent V̇A/Q̇ mismatch with elevated total physiological dead space and possible sympathetic over-excitation may alter central medullary chemoreceptor characteristics in patients with IPF, at least partially explaining elevated exercise V̇E/V̇CO2. Pulmonary microvascular abnormalities may also be a key contributor to the increased dead space and V̇E/V̇CO2 during exercise in IPF. Patients with IPF and mild mechanical restriction have relatively preserved gas transfer between the alveoli and capillaries, even in fibrotic lung regions with interstitial thickening. This suggests that regional capillary hypoperfusion in IPF with mild restriction, despite a relatively preserved alveolar-capillary interface, may lead to V̇A/Q̇ mismatch (specifically an increased proportion of high V̇A/Q̇ lung units), which would increase total physiologic dead space and V̇E/V̇CO2. The relative contribution of increased chemosensitivity and/or pulmonary microvascular abnormalities to elevated exercise V̇E/V̇CO2 in patients mild IPF has not been determined and are the primary focus of this study.

Treatment options for dyspnea management in IPF are limited. Recent work from the INSTAGE trial showed that a combination of nintedanib (anti-fibrotic) and sildenafil (pulmonary vasodilator) showed minimal improvement in dyspnea. However, improvements in physical activity and gas-exchange in patients with IPF following 8-week treatment of inhaled nitric oxide (iNO), a selective pulmonary vasodilator have been demonstrated in other, more recent studies. Since patients with mild forms of IPF are thought to have a relatively intact capillary bed but a relatively high physiological dead space due to attenuation of regional pulmonary perfusion, inhaled selective vasodilation may be more beneficial than in advanced disease with fixed microvascular destruction. This is supported by recent work demonstrating a reduced V̇E/V̇CO2 (reflecting a decrease in physiological dead space) and dyspnea during exercise in patients with mild chronic obstructive pulmonary disease with minimal or no emphysema. Importantly, arterial O2 saturation was normal throughout exercise and unaffected by iNO, which suggests no deleterious effects of iNO on overall gas-exchange. The reduction in V̇E/V̇CO2 during exercise with iNO suggests that iNO increases pulmonary microvascular perfusion heterogeneity, leading to improved V̇A/Q̇ matching, reduced dead space and therefore a lower ventilation for a given metabolic demand.

As an exploratory outcome, we will determine whether iNO improves V̇A/Q̇ and reduces dead space and attendant dyspnea, in patients with IPF and mild mechanical restriction. Moreover, this would clearly establish if partially reversible vascular dysfunction contributes to V̇A/Q̇ mismatch, elevated V̇E/V̇CO2, inspiratory neural drive and dyspnea exists in non-hypoxemic patients with IPF and minimal mechanical abnormalities.

Rationale: It has been well established that patients with advanced IPF have mechanical and pulmonary gas exchange abnormalities which require compensatory increases in inspiratory neural drive and an exaggerated ventilatory response to exercise with consequent increase in activity-related dyspnea. However, very little work has been done to understand mechanisms of exertional dyspnea in patients IPF in whom restrictive mechanics and hypoxemia are not prominent. The proposed work has the potential to not only provide important physiological insight into the underlying mechanisms for increased V̇E/V̇CO2 and inspiratory neural drive, but also to examine therapeutic avenues to improve ventilatory efficiency, dyspnea, exercise capacity and ultimately quality of life in patients with IPF.

ELIGIBILITY:
Inclusion criteria:

* clinically stable, as defined by stable hemodynamic status, optimized medical treatment, no changes in medication dosage or frequency of administration with no hospital admissions in the preceding 6 weeks;
* Mild or absent mechanical restriction as determined by a total lung capacity (TLC) >70% predicted;
* male or female non-pregnant adults >40 years of age;
* ability to perform all study procedures and provide informed consent.
* A key IPF inclusion criterion includes, in addition to the above, a clinical diagnosis of idiopathic pulmonary fibrosis.

Exclusion criteria:

* women of childbearing potential who are pregnant or trying to become pregnant;
* computed tomography evidence of any (significant) emphysema
* evidence of airway obstruction (forced expiratory volume in 1 s/forced vital capacity <0.70,
* active cardiopulmonary disease (other than IPF) or other comorbidities that could contribute to dyspnea and exercise limitation;
* history/clinical evidence of asthma, atopy and/or nasal polyps;
* currently taking phosphodiesterase type 5 inhibitors;
* important contraindications to clinical exercise testing, including inability to exercise because of neuromuscular or musculoskeletal disease(s);
* body mass index (BMI) <18.5 or ≥35.0 kg/m2;
* use of daytime oxygen or exercise-induced O2 desaturation (<80% on room air).

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-04-21 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Ventilatory efficiency (VE/VCO2) | During exercise test on visit 4 and 5, every 1 minute, through end-exercise (average time 6-10minutes).
  Ventilatory efficiency will be measured by expired gas analysis. Measurements will be collected on a breath-by breath basis and compared with predicted values based on age and height. Three main time points will be evaluated: "rest" will be defined as the steady-state period after at least 3 minutes of breathing on the mouthpiece before exercise starts; "isotime" will be defined as the last 30-sec increment of each minute (i.e. 1-min, 2-min, 3-min) during the incremental exercise test and at 2 minutes (or the longest time achieved by all subjects) during the constant load exercise tests, and; "end-exercise" will be defined as the last 30-sec of loaded pedaling.
Inspiratory Neural Drive (IND) as measured by Diaphragmatic electromyography (EMGdi) | During exercise test on visit 4 and 5, every 1 minute, through end-exercise (average time 6-10minutes).
  An esophageal electrode-balloon catheter consisting of 5 electrode pairs and two balloons, will be inserted nasally and positioned for optimal recoding. Electromyogram output of the diaphragm (used as an index of inspiratory neural drive to crural diaphragm or diaphragm activation; EMGdi) will be recorded continuously at rest and during exercise. Maximal EMGdi (EMGdi,max) will be determined from inspiratory capacity (IC) maneuvers. EMGdi/EMGdi,max will be used as an index of the inspiratory neural drive to the crural diaphragm.

SECONDARY OUTCOMES:
Dyspnea Intensity | During exercise test on visit 4 and 5, every 1 minute, through end-exercise (average time 6-10minutes).
  Dyspnea (respiratory discomfort) will be defined as the "sensation of breathing discomfort" experienced at rest and during pedaling. Measurements will be made at rest (the steady-state period after at least 3 minutes of breathing on the mouthpiece before exercise starts), at two-minute intervals during exercise, and at end-exercise (at 2 minutes or the last 30-sec of loaded pedaling achieved by all the participants). The intensity (strength) of sensations will be rated using the modified 10-point Borg scale.

CONTACTS AND LOCATIONS:
Overall Officials: Denis E O'Donnell, MD, Principal Investigator — Principal Investigator, Professor
Locations (1):
- Respiratory Investigation Unit, Kingston General Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Milne KM, Ibrahim-Masthan M, Scheeren RE, James MD, Phillips DB, Moran-Mendoza O, Ja N, O'Donnell DE. Inspiratory neural drive and dyspnea in interstitial lung disease: Effect of inhaled fentanyl. Respir Physiol Neurobiol. 2020 Nov;282:103511. doi: 10.1016/j.resp.2020.103511. Epub 2020 Aug 3. PMID 32758677
- [Background] Faisal A, Alghamdi BJ, Ciavaglia CE, Elbehairy AF, Webb KA, Ora J, Neder JA, O'Donnell DE. Common Mechanisms of Dyspnea in Chronic Interstitial and Obstructive Lung Disorders. Am J Respir Crit Care Med. 2016 Feb 1;193(3):299-309. doi: 10.1164/rccm.201504-0841OC. PMID 26407036
- [Background] Farina S, Bruno N, Agalbato C, Contini M, Cassandro R, Elia D, Harari S, Agostoni P. Physiological insights of exercise hyperventilation in arterial and chronic thromboembolic pulmonary hypertension. Int J Cardiol. 2018 May 15;259:178-182. doi: 10.1016/j.ijcard.2017.11.023. PMID 29579597
- [Background] Kolb M, Raghu G, Wells AU, Behr J, Richeldi L, Schinzel B, Quaresma M, Stowasser S, Martinez FJ; INSTAGE Investigators. Nintedanib plus Sildenafil in Patients with Idiopathic Pulmonary Fibrosis. N Engl J Med. 2018 Nov 1;379(18):1722-1731. doi: 10.1056/NEJMoa1811737. Epub 2018 Sep 15. PMID 30220235
- [Background] Nathan SD, Flaherty KR, Glassberg MK, Raghu G, Swigris J, Alvarez R, Ettinger N, Loyd J, Fernandes P, Gillies H, Kim B, Shah P, Lancaster L. A Randomized, Double-Blind, Placebo-Controlled Study of Pulsed, Inhaled Nitric Oxide in Subjects at Risk of Pulmonary Hypertension Associated With Pulmonary Fibrosis. Chest. 2020 Aug;158(2):637-645. doi: 10.1016/j.chest.2020.02.016. Epub 2020 Feb 21. PMID 32092321
- [Background] Phillips DB, Brotto AR, Ross BA, Bryan TL, Wong EYL, Meah VL, Fuhr DP, van Diepen S, Stickland MK; Canadian Respiratory Research Network. Inhaled nitric oxide improves ventilatory efficiency and exercise capacity in patients with mild COPD: A randomized-control cross-over trial. J Physiol. 2021 Mar;599(5):1665-1683. doi: 10.1113/JP280913. Epub 2021 Jan 25. PMID 33428233